CLINICAL TRIAL: NCT05308199
Title: Comparison of Thoracic Manipulation & MET for Chronic Mechanical Neckache; a Single Blinded Clinical Trail
Brief Title: Physiotherapy Techniques in Adult Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Muhammad salman, PT, Principal researcher, Neuro Counsel Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2022-03-18; First posted 2022-04-01 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Neckache
Keywords: neckache
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: 2 groups , geoup A named as control group and group B named as experimental group
Masking Description: participants didn't know in which group they are and what type of treatment they are given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): thoracic manipulation group
  Interventions: Other: thoracic manipulation
- control (Active Comparator): MET group
  Interventions: Other: muscle enegy technique

INTERVENTIONS:
Other: thoracic manipulation — thoracic manipulation for unlocking of facet joints
  Arms: experimental
Other: muscle enegy technique — to release muscle spasm of cervical musces
  Arms: control

SUMMARY:
To compare the effectiveness of thoracic manipulation and MET on chronic mechanical neckache

DETAILED DESCRIPTION:
it is a randomized control clinical trail to compare the effectiveness of physical exercises for the management of chronical mechanical neckache .so we employed thoracic manipulation for experimental group and MET (muscle energy technique) for control group

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with mechanical neck pain having age group of 18 to 60 years.
* Mechanical neck pain having activities of daily living
* Mechanical Neck pain affecting sleep

Exclusion Criteria:

Patients with following conditions will be excluded

* Osteoporosis
* Radiculopathy
* Pregnancy
* Systemic inflammatory condition
* Neurological deficit
* Arthritic conditions
* Head injuries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 6 weeks
  MINIMUM MEANS NO PAIN AND MAXIMUM SCORE MEANS WORST PAIN

SECONDARY OUTCOMES:
frequency of pain | 6 week
  MINIMUM MEANS NO PAIN AND MAXIMUM SCORE MEANS WORST PAIN

OTHER OUTCOMES:
duration of pain | 6 weeks
  MINIMUM MEANS NO PAIN AND MAXIMUM SCORE MEANS WORST PAIN

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD SALMAN, M.Phil*, Principal Investigator — the neurocouncil hospital
Locations (2):
- Pakistan (2):
  - Muhammad Salman, Islamabad, Fedral
  - the Neurocouncil Clinic, Islamabad, Fedral

REFERENCES:
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284